CLINICAL TRIAL: NCT06840574
Title: The Effect of Nutritional Supplementation on Actinic Purpura: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SP0022 Cyruta Plus
Record Dates: First submitted 2025-02-06; First posted 2025-02-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Skin Health; Skin Aging of Face and Hands; Healthy; Ecchymosis
MeSH Terms: conditions — Ecchymosis | interventions — Honey; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cyruta Plus (Experimental): Total of 27 mg daily
  Interventions: Dietary Supplement: Cyruta Plus: A Whole-Food Based Vitamin C supplement containing organic buckwheat (aerial parts) juice powder, organic buckwheat flour, bovine adrenal Cytosol™ extract, oat flour, honey, ascorbic acid
- Low-dose Vitamin C (Active Comparator): Total of 27 mg daily
  Interventions: Dietary Supplement: Low Dose Vitamin C
- High-dose Vitamin C (Active Comparator): Total of 500 mg daily
  Interventions: Dietary Supplement: High Dose Vitamin C

INTERVENTIONS:
Dietary Supplement: Cyruta Plus: A Whole-Food Based Vitamin C supplement containing organic buckwheat (aerial parts) juice powder, organic buckwheat flour, bovine adrenal Cytosol™ extract, oat flour, honey, ascorbic acid — 27 mg vitamin C, organic buckwheat (aerial parts) juice powder, organic buckwheat flour, bovine adrenal Cytosol™ extract, oat flour, honey, ascorbic acid, and calcium stearate
  Arms: Cyruta Plus
Dietary Supplement: Low Dose Vitamin C — 27 mg ascorbic acid
  Arms: Low-dose Vitamin C
Dietary Supplement: High Dose Vitamin C — 500 mg ascorbic acid
  Arms: High-dose Vitamin C

SUMMARY:
Purpura is a macule or papule of blood in the skin. It is mostly seen in mature skin that is often prone to significant bruising. Small lesions of less than 5 mm are called petechiae and larger ones, found mostly in subcutaneous tissue, are called ecchymosis. Actinic purpura occurs almost exclusively in elderly populations. This single-blind randomized clinical trial evaluates the effect of an 8-week nutritional supplement intervention in comparison with isolated vitamin C supplements on actinic purpura in older adults. We will enroll thirty (30) otherwise healthy participants, both male and female, aged 55 years and older. Changes in participants' skin condition will be assessed at visit 1 (baseline), visit 2 (4-week), and visit 3 (8-week) using questionnaires, standard digital photography, and clinical grading of the skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals aged ≥ 55 years old.
* Self-reported having actinic purpura lesions at the time of enrollment or a history of actinic purpura lesions.
* Self-reported not using prescription or over-the-counter products that contain aluminum, iron, proton pump inhibitors (PPIs), and/or topical retinol (used locally in areas of bruising).
* If on a chronic medication that does not result in exclusion, participant must self-report being on a stable dose for the last 3 months prior to the start of the trial.
* Able and willing to read and voluntarily sign the study Informed Consent Form (ICF).
* Able and willing to comply with study protocol and all study-related guidelines.
* Not concomitantly participating in a study involving nutritional products.

Exclusion Criteria:

* Not complying with the study protocol.
* Having a known allergy or intolerance to nuts, seeds, fruits, vegetables, oils, and fish.
* Having a known allergy, intolerance, or dietary restriction to any of the study ingredients (Vitamin C, organic buckwheat (aerial parts) juice powder, organic buckwheat flour, bovine adrenal Cytosol™ extract, oat flour, honey, ascorbic acid, and calcium stearate).
* Having a clinically significant condition that is severe, progressive, or uncontrolled and would compromise the study or their well-being or would prevent the participant from meeting or performing study requirements. This includes but is not limited to dysphagia (or difficulty swallowing), liver or kidney disease, bone marrow problems, Ehlers-Danlos syndrome, lupus, alcohol misuse, cancer, or HIV and other infections.
* Having active dermatological conditions. Patients with active, severe skin conditions that might interfere with the study's conduct or outcomes including widespread psoriasis, untreated chronic skin ulcers, or other severe dermatological disorders.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 8 weeks
  The number of participants who report a reduction in the number of purpura lesions as evaluated through dermatological examination before and after supplementation.

SECONDARY OUTCOMES:
Secondary Endpoint | 8 weeks
  Average decrease in actinic purpura lesion measurements in millimeters across participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Standard Process - Nutrition Innovation Center, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No